CLINICAL TRIAL: NCT06357052
Title: The Study of Lithogenesis Processes in Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Acronym: LINA
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 2701
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: NAFLD; Urinary Lithiasis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NAFLD patients without liver cirrhosis (NLCs, n = 28)
- NAFLD patients with liver cirrhosis (LCs, n = 14)
- healthy individuals (HIs, n = 12)

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is the most common cause of chronic liver disease, ranging from pure steatosis to non-alcoholic steatohepatitis and ultimately to liver cirrhosis. In order to study the association between NAFLD and nephrolithiasis while minimizing the confounding effect of metabolic syndrome, we investigated the impact of different degrees of NAFLD severity on potential risk factors for stone formation.

ELIGIBILITY:
Inclusion Criteria:

* subject >= 18 years old
* able to sign the ICF
* Liver biopsy with report compatible with NAFLD

Exclusion Criteria:

* alchol use > 20g/die
* other causes of liver disease
* active neoplasm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 subjects suffering from NAFLD histologically ascertained by routine liver biopsy performed at the P.O. liver surgeries Columbus relating to the Gastroenterology Area Units.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
the analysis of the correlation between the degree of severity of NAFLD And urinary lithogenic profilecharacterized by reduced urinary magnesium and altered urinary ammonium excretion. | 15 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico A.Gemelli IRCCS, Roma, Italy